CLINICAL TRIAL: NCT06382493
Title: Efficacy of Tegoprazan-containing Sequential Therapy Compared to Proton Pump Inhibitor-based Eradication in South Korea, a Region With High Antimicrobial Resistance: A Prospective Randomized Single Tertiary Center Study
Brief Title: Tegoprazan-containing Sequential for H. Pylori
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2011-648-005
Record Dates: First submitted 2024-04-20; First posted 2024-04-24 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esomeprazole-containing sequential H. pylori eradication therapy (conventional method) (Active Comparator): esomeprazole (40 mg) plus amoxicillin (1000 mg) twice a day for initial 5 days, and then esomeprazole (40 mg) with clarithromycin (500 mg) and metronidazole (500 mg) twice a day for the remaining 5 days.
  Interventions: Drug: Esomeprazole-containing sequential H. pylori eradication therapy
- Tegoprazan-containing sequential H. pylori eradication therapy (experimental method) (Experimental): tegoprazan (50 mg) plus amoxicillin (1000 mg) twice a day for initial 5 days, and then tegoprazan (50 mg) with clarithromycin (500 mg) and metronidazole (500 mg) twice a day for the remaining 5 days.
  Interventions: Drug: Tegoprazan-containing sequential H. pylori eradication therapy

INTERVENTIONS:
Drug: Tegoprazan-containing sequential H. pylori eradication therapy — tegoprazan was administered, instead propton-pump inhibitor, as acid blockade in H. pylori eradication sequential therapy
  Arms: Tegoprazan-containing sequential H. pylori eradication therapy (experimental method)
Drug: Esomeprazole-containing sequential H. pylori eradication therapy — Esomeprazole was administered as acid blockade in H. pylori eradication sequential therapy (conventional acid blockade method for sequential eradication therapy)
  Arms: Esomeprazole-containing sequential H. pylori eradication therapy (conventional method)

SUMMARY:
As H. pylori eradication, the investigators prepared a randomized controlled clinical trial whether tegoprazan-containing 10-day sequential treatment was effective compared to conventional PPI-containing 10-day sequential eradication therapy

DETAILED DESCRIPTION:
Eradication treatment containing potassium-competitive acid blocker has shown acceptable eradication efficacy. In regions such as Korea, where the prevalence of antimicrobial resistance is high, alternative combinations of antibiotics such as sequential or concomitant therapy are needed. This study compared the outcome of sequential therapy containing tegoprazan, a new potassium-competitive acid blocker, with the conventional esomeprazole-containing sequential therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients who had H. pylori infection proved by positive test result of urea breath test (UBT), rapid urase test or pathologic examination (warthin-giemsa staining)

Exclusion Criteria:

* congestive heart failure, NYHA III or IV
* end-stage renal disease
* alcoholics
* drug abusers
* pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 2 or 3 month
  Efficacy of H. pylori eradication therapy. confirmed by negative UBT test

SECONDARY OUTCOMES:
Adverse events | up to 6 month
  any adverse events occured during or after intervention (eradication therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, Prof., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JW, Kim N, Lee J, Jo SY, Lee DH. Efficacy of Tegoprazan-Containing Sequential Eradication Treatment Compared to Esomeprazole-Containing Sequential Eradication of Helicobacter pylori in South Korea, a Region With High Antimicrobial Resistance: A Prospective, Randomized, Single Tertiary Center Study. Helicobacter. 2024 Sep-Oct;29(5):e13143. doi: 10.1111/hel.13143. PMID 39434634